CLINICAL TRIAL: NCT03670589
Title: Vestibular Evaluation Before and After Treatment of Vestibular Schwannoma. Comparison of Gamma Knife Radiosurgery and Microsurgical Resection
Brief Title: Vestibular Evaluation After Vestibular Schwannoma Treatment
Acronym: EVTSVCGEC
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, EssaiClinique_EVTSVCGEC, Vestibular Evaluation Before and After Treatment of Vestibular Schwannoma. Comparison of Gamma Knife Radiosurgery and Microsurgical Resection., University Hospital, Grenoble
Other Study IDs: 38RC18.098; 2018-A01208-47 (Other: ID RCB)
Record Dates: First submitted 2018-08-24; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Dizziness
Keywords: vestibular schwannoma; gammaknife radiosurgery; vestibular evaluation
MeSH Terms: conditions — Dizziness; Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- radiosurgery gammaknife group: Patient treated by radiosurgery gammaknife for a one side vestibular schwannoma
  Interventions: Radiation: Radiosurgery gammaknife
- microsurgery resection group: Patient treated by microsurgery resection for a one side vestibular schwannoma
  Interventions: Procedure: Microsurgery resection

INTERVENTIONS:
Radiation: Radiosurgery gammaknife — This procedure use intense gamma ray, which are concentrated to the precise volume of the tumor that used to stop the progression of the tumor
  Groups: radiosurgery gammaknife group
Procedure: Microsurgery resection — Classical surgical approach with oto-neurosurgery procedures
  Groups: microsurgery resection group

SUMMARY:
Vestibular schwannoma is a benign tumor located on the vestibular nerve. Patient could present dizziness symptoms cause to the tumor, and at least after the treatment by gamaknife radiosurgery or microsurgery resection.

Only few studies keep the interest about dizziness symptoms and treatment modality in vestibular schwannoma.

In the study dizziness symptoms were compared before and after the treatment of vestibular schwannoma by radiosurgery gammaknife or microsurgery resection. 2 scales were used : dizziness handicap inventory (DHI) and dizziness functionnal scale (AAO).

ELIGIBILITY:
Inclusion Criteria:

* patient treated of an one side vestibular schwannoma between 01/01/2012 and 31/12/2017, follow at the Grenoble University Hospital
* treatment : gamaknife radiosurgery or microsurgery resection
* no opposition of the patient

Exclusion Criteria:

* association of gamaknife radiosurgery and microsurgery resection
* bilateral vestibular schwannoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The popultaion include patients treated by gamaknife radiosurgery or microsurgery resection for a one side vestibular schwannoma between 01/01/2012 and 31/12/2017, follow at the Grenoble University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Vestibular evaluation DHI | From 4 years to 6 months
  The investigator use a standarised scale :
  - Dizziness Handicap Inventory (DHI). This scale combines 25 questions with three answers for each proposition about dizzyness in daily life situation : everytime (quote 4), sometimes (quote 2), never (quote 0). The scores are summing to obtain a value on 100.
  The scale is completed before and after the treatement. The investigator send the scale to the patient by mail way.
Vestibular evaluation AAO | From 4 years to 6 months
  The investigator use a standarised scale :
  - Dizziness Functionnal Scale (AAO), this is a scale quote from 1 (no symptoms of dizzyness) to 6 (major disability). The patient have to choise only one item that correspond to the condition.
  The scale is completed before and after the treatement. The investigator send the scale to the patient by mail way.

SECONDARY OUTCOMES:
Facial fonction | From 4 years to 6 months
  House and Brackmann scale :
  This scale is a standarised assessment of facial fonction from grade I : normal ; to grade VI : total paralysis.
  Each scale is completed after the treatement.
Hearing function | From 4 years to 6 months
  This information is based on a question to the patient about the usefulness of hearing prothesis.
  So there are 2 groups : useful hearing (normal hearing or used hearing prothesis) or useless hearing (unsused hearing prothesis)
  The information is completed before and after the treatement.
Tumor control | From 4 years to 6 months
  Tumor control is based on MRI size description (in mm):
  So there are 2 groups : controled or evolution of the tumor.
  * for microsurgery resection group the investigator keeps interest about the remaining size
  * for radiosurgery gammaknife group the investigator keeps interest about the stability or the reduction of the tumor
  The result is completed after the treatement.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlson ML, Tveiten OV, Driscoll CL, Neff BA, Shepard NT, Eggers SD, Staab JP, Tombers NM, Goplen FK, Lund-Johansen M, Link MJ. Long-term dizziness handicap in patients with vestibular schwannoma: a multicenter cross-sectional study. Otolaryngol Head Neck Surg. 2014 Dec;151(6):1028-37. doi: 10.1177/0194599814551132. Epub 2014 Oct 1. PMID 25273693
- [Background] Park CE, Park BJ, Lim YJ, Yeo SG. Functional outcomes in retrosigmoid approach microsurgery and gamma knife stereotactic radiosurgery in vestibular schwannoma. Eur Arch Otorhinolaryngol. 2011 Jul;268(7):955-9. doi: 10.1007/s00405-011-1596-9. Epub 2011 Apr 11. PMID 21479879
- [Background] Pollock BE, Driscoll CL, Foote RL, Link MJ, Gorman DA, Bauch CD, Mandrekar JN, Krecke KN, Johnson CH. Patient outcomes after vestibular schwannoma management: a prospective comparison of microsurgical resection and stereotactic radiosurgery. Neurosurgery. 2006 Jul;59(1):77-85; discussion 77-85. doi: 10.1227/01.NEU.0000219217.14930.14. PMID 16823303
- [Background] Coelho DH, Roland JT Jr, Rush SA, Narayana A, St Clair E, Chung W, Golfinos JG. Small vestibular schwannomas with no hearing: comparison of functional outcomes in stereotactic radiosurgery and microsurgery. Laryngoscope. 2008 Nov;118(11):1909-16. doi: 10.1097/MLG.0b013e31818226cb. PMID 18849856